CLINICAL TRIAL: NCT02767752
Title: A Single Center, Randomized, Double-Blind, Placebo-Controlled Phase 2 Study of Gemcitabine (GEM) and Capecitabine (CAP) With or Without T-ChOS as Adjuvant Therapy in Patients With Surgically Resected Pancreatic Cancer.
Brief Title: Gemcitabine and Capecitabine With or Without T-ChOS as Adjuvant Therapy for Patients With Resected Pancreatic Cancer
Acronym: CHIPAC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual and change of SOC (FOLFIRINOX in adjuvant setting)
Sponsor: Herlev Hospital (Other)
Collaborators: GENIS (Unknown)
Responsible Party: Principal Investigator, Inna Chen, MD, Staff specialist, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GI 1604
Record Dates: First submitted 2016-05-06; First posted 2016-05-10 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Pancreatic Cancer
Keywords: Resectable pancreatic cancer; Adjuvant
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Sugars; Capecitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- T-ChOS + Gemcitabine + Capecitabine (Experimental): T-ChOS: 600 mg given p.o. (two capsules, each 300 mg) daily in the morning 30 minutes before food.
  Gemcitabine: 1000 mg/m²i.v. on day 1, day 8 and day 15 of every 28 day cycle. Capecitabine: 1660 mg/m²/day p.o. twice daily 21/28 day i. e. 24 weeks.
  Interventions: Dietary Supplement: T-ChOS; Drug: Gemcitabine; Drug: Capecitabine
- Placebo + Gemcitabine + Capecitabine (Placebo Comparator): Placebo: 600 mg given p.o. (two capsules, each 300 mg) daily in the morning 30 minutes before food.
  Gemcitabine: 1000 mg/m²i.v. on day 1, day 8 and day 15 of every 28 day cycle. Capecitabine: 1660 mg/m²/day p.o. twice daily 21/28 day i. e. 24 weeks.
  Interventions: Drug: Gemcitabine; Dietary Supplement: Placebo; Drug: Capecitabine

INTERVENTIONS:
Dietary Supplement: T-ChOS
  Other Names: Benecta™
  Arms: T-ChOS + Gemcitabine + Capecitabine
Drug: Gemcitabine
Dietary Supplement: Placebo
  Other Names: Sugar pill manufactured to mimic 300 mg capsule
  Arms: Placebo + Gemcitabine + Capecitabine
Drug: Capecitabine
  Other Names: Xeloda

SUMMARY:
This is a single center, randomized, double-blind, placebo-controlled phase II trial that will compare the efficacy of T-ChOS in combination with gemcitabine to gemcitabine alone as adjuvant treatment for 6 months in patients with surgically resected pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Histologically confirmed resected ductal pancreatic adenocarcinoma with macroscopic complete resection (R0 and R1). Subjects with neuroendocrine (and mixed type) tumors are excluded
3. Subject should be able to start treatment no later than 12 weeks post-surgery
4. Male or non-pregnant, non-lactating females who are ≥18 years of age at the time of signing the informed consent form (ICF)
5. ECOG/WHO Performance Status (PS) 0-1
6. Females of child-bearing potential (defined as a sexually mature woman who (1) has not undergone hysterectomy [the surgical removal of the uterus] or bilateral oophorectomy [the surgical removal of both ovaries] or (2) has not been naturally postmenopausal for at least 24 consecutive months [i.e., has had menses at any time during the preceding 24 consecutive months]) must:

   * Agree to the use of two physician-approved contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) while on study IP; and for 3months following the last dose of IP
   * Has negative serum pregnancy test (β-hCG) result at screening
7. Male subjects:

   • Must practice true abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for 6 months following IP discontinuation, even if he has undergone a successful vasectomy
8. Understand and voluntarily sign an ICF prior to any study related assessments or procedures being conducted
9. Be able to adhere to the study visit schedule and other protocol requirements
10. Acceptable hematology parameters defined as:

    * Absolute neutrophil count (ANC) ≥ 1.5 x 10⁹/L
    * Platelet count ≥ 100 x 10⁹/L
    * Haemoglobin ≥ 5.6 mmol/L
11. Acceptable liver function defined as:

    * Serum bilirubin < 1.5 x upper limit of normal (ULN)
    * ASAT/ALAT < 2.5 x ULN
12. Acceptable renal function with a creatinine clearance ≥ 50 mL/min/ (e.g., using the Cockroft-Gault formula)

Exclusion Criteria:

1. Prior neo-adjuvant treatment, radiation therapy, or systemic therapy for pancreatic adenocarcinoma
2. Presence of or history of metastatic or locally recurrent pancreatic adenocarcinoma
3. Other malignancies, except adequately treated basal carcinoma or squamous cell carcinoma of the skin or in situ cervix carcinoma or incidental prostate cancer (T1a, Gleason score ≤ 6, PSA < 0.5 ng/ml), or any other tumor with a DSF survival of ≥ 5 years
4. History of serious or concurrent illness or uncontrolled medical disorder; any medical condition that might be aggravated by chemotherapy treatment or which could not be controlled; including, but not restricted to:

   * Active infection requiring antibiotics within 2 weeks before the study inclusion
   * Concurrent congestive heart failure NYHA class III - IV
   * Unstable angina pectoris, or myocardial infarction within 6 months and/or prior poorly controlled hypertension
   * History of interstitial lung disease, slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis or multiple allergies
   * Concomitant use of immunosuppressive or myelosuppressive medications that would in the opinion of the investigator, increase the risk of serious neutropenic complications
5. Known or suspected allergy to the investigational agents or any agents given in association with this trial
6. Any psychological, familial, sociological, or geographical condition which does not permit protocol compliance and medical follow-up
7. Enrollment in any other clinical protocol or investigational study with an interventional agent or assessments that may interfere with study procedures
8. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study
9. Any condition that confounds the ability to interpret data from the study
10. Unwillingness or inability to comply with study procedures
11. Current use of anticoagulation therapy such as heparins both unfractionated and low molecular weighted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | up to approximately 9 months
  Time from the date of randomization to the date of disease recurrence or death, whichever is earlier.

SECONDARY OUTCOMES:
Overall Survival | up to approximately 18 months
  Time from the date of randomization to the date of death
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to approximately 18 months
  Assesment by CTCAE v4.0
Quality of Life | up to approximately 18 months
  Quality of Life Questionnaire C30 (QLQ-C30) Version 3.0

OTHER OUTCOMES:
Determination of plasma YKL-40 | up to approximately 9 months
  Measurement using an enzyme linked-immunosorbent assay
Determination of plasma IL-6 | up to approximately 9 months
  Measurement using an enzyme linked-immunosorbent assay

CONTACTS AND LOCATIONS:
Overall Officials: Inna Chen, MD, Principal Investigator — Herlev & Gentofte Hospital
Locations (1):
- Department of Oncology, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: Yes